CLINICAL TRIAL: NCT05483582
Title: Clinical Trial to Evaluate the Efficacy and Safety of a 4-channel Swallowing Function Electrical Stimulation Device Compared to a 2-channel Swallowing Function Electrical Stimulation Device for the Rehabilitation Mechanism
Brief Title: Clinical Trial for Clinical Excellence and Safety Evaluation of 4-channel Functional Electric Stimulator
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-2103-672-001
Record Dates: First submitted 2021-11-01; First posted 2022-08-02 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classical electrical stimulation protocol (control group) (Active Comparator): * Apply 2-channel electrical stimulation device with protocol 1.
  * It will simultaneously stimulate bilateral suprahyoid, bilateral thyrohyoid muscle with 2-channel electrical stimulation device.
  * Basic intervention involves 600-900 minutes of electrical stimulation for 2 weeks. (based on 60 minutes per 1 time, applied 10 times(+5 times, within 1 week))
  * With the consent of the patient, an additional evaluation is performed after additional 2 weeks of intervention, which is use as an exploratory indicator.
  * After application of the device, we evaluate videofluoroscopic swallowing study(VFSS) for evaluation of swallowing function.
  * In addition, we evaluate clinical questionnaires(FOIS, MDADI, Likert scale), nutritional status assessments(MNA-SF), and oral intake assessments.
  * Also, we measure tongue strength through IOPI and body composition changes through Inbody.
  Interventions: Device: 2-channel Electrical Stimulation Device
- revised sequential activation protocol (experimental group) (Experimental): * Apply 4-channel electrical stimulation device with protocol 2.
  * It sequentially stimulates bilateral suprahyoid muscle(ch 1, ch 2), bilateral thyrohyoid muscle(ch 3), bilateral sternothyroid muscle(ch 4) with 4-channel electrical stimulation device.
  * Basic intervention involves 600-900 minutes of electrical stimulation for 2 weeks. (based on 60 minutes per 1 time, applied 10 times(+5 times, within 1 week))
  * With the consent of the patient, an additional evaluation is performed after additional 2 weeks of intervention, which is use as an exploratory indicator.
  * After application of the device, we evaluate videofluoroscopic swallowing study(VFSS) for evaluation of swallowing function.
  * In addition, we evaluate clinical questionnaires(FOIS, MDADI, Likert scale), nutritional status assessments(MNA-SF), and oral intake assessments.
  * Also, we measure tongue strength through IOPI and body composition changes through Inbody.
  Interventions: Device: 4-channel Electrical Stimulation Device

INTERVENTIONS:
Device: 4-channel Electrical Stimulation Device — electrical stimulation at muscles which related with deglutition
  Arms: revised sequential activation protocol (experimental group)
Device: 2-channel Electrical Stimulation Device — electrical stimulation at muscles which related with deglutition
  Arms: classical electrical stimulation protocol (control group)

SUMMARY:
This study is a pilot study to prepare clinical trials to evaluate the safety and effectiveness of 4-channel electric stimulation therapy devices as a newly developed function for the treatment of dysphagia disorders.

The purpose of this study is to investigate the difference in effect by the electric stimulation method and to obtain the values such as mean, standard deviation and so on, and to determine the number of subjects to be studied for clinical trials of validation permission in the future.

DETAILED DESCRIPTION:
* Design: Prospective study
* Inclusion criteria of patient group: who has a dysphagia symptom and confirmed by video-fluoroscopic swallowing study
* Intervention: Participants are divided into two group and applied electrical stimulation by a "Synchronized Electrical Stimulation Device(SESD)" in different protocol
* Main outcome measures: Videofluoroscopic Dysphagia Scale (VDS), Penetration aspiration scale (PAS), Measured by kinematic metaphysical analysis. The dietary status of the subjects was evaluated by the Functional Oral Intake Scale (FOIS), and the M.D Anderson dysphagia inventory was used to measure the diet-related quality of life. The Likert scale is used to evaluate the satisfaction with the application of the electric stimulation therapy device of the study subjects.
* Secondary outcome measures: Verifying the safety of functional electric stimulation therapy device for dysphagia, measuring the effect on Tongue Strength through IOPI, the effect on changes in body composition through Bioelectrical Impedance Analysis (BIA; InBody S10, InBody, Inc.), and whether there is a significant change in actual patient intake and nutritional status through oral intake survey and MNA-SF measure. An exploratory comparison of intervention effects over time between 2-week and 4-week interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with oropharyngeal dysphagia confirmed by video fluoroscopy
* Patients with oropharyngeal dysphagia due to central nervous system disease who clinically require application of an electrical stimulation treatment device for dysphagia
* Patients aged between 19 and under 90 years of age regardless of gender
* Those who voluntarily consent to the clinical trial and can visit for the next observation
* Patients with dysphagia within 6 months (including patients with dysphagia due to stroke, traumatic brain injury, cervical spine injury, etc.)

Exclusion Criteria:

* In case of refusal of inspection
* Who do not agree
* When instructions cannot be performed due to mental illness, etc.
* Those who have dysphagia due to respiratory failure, cervical spine surgery, head and neck surgery, and chemotherapy and radiation treatment of the neck
* Pregnant and lactating women
* Pre-interview is conducted only with women of childbearing age to determine whether they are pregnant or lactating. If pregnancy is confirmed during the pre-interview, it is excluded from the test.
* Patients who cannot apply electrical stimulation therapy due to allergies or hypersensitivity reactions
* Others who have comorbidities (e.g., malignant tumors, severe renal/liver/lung diseases, blood clotting abnormalities, etc.) that are inappropriate for participation in clinical trials as judged by the researcher
* Persons with pacemakers and other internal electrical stimulators
* Those who are participating in other clinical trials at the time of screening
* Those who are judged by other researchers to be inappropriate for this clinical trial

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of VDS total change | 300 to 600 minutes
  Comparison of VDS total change between the two groups using the results of the video fluoroscopic swallowing test between the experimental group and the control group

SECONDARY OUTCOMES:
Using the results of the video fluoroscopic swallowing test | 300 to 600 minutes
  Comparison of changes in VDS (oral score, pharyngeal score), PAS (Penetration Aspiration Scale) and kinematic analysis using the results of video fluoroscopic swallowing test.
Results of pre- and post-intervention surveys | 30 to 60 minutes
  The dietary status of the subjects was evaluated by the Functional Oral Intake Scale (FOIS), and the M.D anderson dysphagia inventory was used to measure the diet-related quality of life.
Satisfaction evaluation of treatment device | 10 to 30 minutes
  The Likert scale is used to evaluate the satisfaction with the application of the electric stimulation therapy device of the study subjects.
Exploratory observation of the effect of electrical stimulation therapy | 30 to 60 minutes
  Exploratory observation of the effect of electrical stimulation therapy on tongue strength through IOPI, comparison of fluctuation values of body composition through Bioelectrical Impendance Analysis (BIA; InBody), measurement of changes in oral intake and malnutrition index before and after intervention and MNA-SF questionnaire do.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Medicine, Seoul National University Bundang Hospital, Seoul National University College of Medicine, Seongnam-si, Gyeonggi-do, South Korea